CLINICAL TRIAL: NCT01300351
Title: A Randomised, Double-Blind, Parallel-Group, Multicentre Study Comparing the Efficacy and Tolerability of Fulvestrant 500 mg Versus 250 mg in Postmenopausal Women With ER+ Advanced Breast Cancer Progressing or Relapsing After Previous Endocrine Therapy
Brief Title: Comparing the Efficacy and Tolerability of Fulvestrant 500 mg Versus 250 mg in Advanced Breast Cancer Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D6997L00021
Record Dates: First submitted 2011-02-17; First posted 2011-02-21 (Estimated); Results first posted 2015-04-24 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Breast Cancer
Keywords: Advanced breast cancer; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fulvestrant 500mg (Experimental): Fulvestrant 500mg (2 syringes of Fulvestrant 250mg), Fulvestrant 500 mg i.m. every 28 (+/- 3) days plus an additional 500 mg on day 14 (+/-3) of first month only
  Interventions: Drug: Fulvestrant
- Fulvestrant 250mg (Active Comparator): Fulvestrant 250mg (1 syringe of fulvestrant 250mg + 1 syringe matching placebo), Fulvestrant 250 mg and matching placebo i.m. every 28 (+/- 3) days plus an additional 2 placebo syringes on day 14 (+/-3) of first month only
  Interventions: Drug: Fulvestrant; Drug: Placebo

INTERVENTIONS:
Drug: Fulvestrant — Fulvestrant was supplied as a castor oil based solution in clear neutral glass pre-filled syringes. Each syringe will contain 250 mg of fulvestrant in 5 ml.
  Other Names: Faslodex
Drug: Placebo — Matching placebo was supplied as a castor oil based solution in clear neutral glass prefilled syringes. Each syringe will contain 5 ml.
  Arms: Fulvestrant 250mg

SUMMARY:
The purpose of this study is to evaluate the efficacy of a new dose of 500mg Fulvestrant with the standard dose of 250mg in Chinese postmenopausal women with oestrogen receptor positive advanced breast cancer who have failed a prior endocrine treatment.

DETAILED DESCRIPTION:
Fulvestrant, at a dose of 250mg every 28 days, is the first oestrogen receptor antagonist with no agonist effects shown to be at least as effective for both TTP (Time to Progression) and OR (Objective Response) as a third-generation aromatase inhibitor in the second-line treatment of advanced breast cancer (Howell et al 2002, Osborne CK et al 2002).In these studies overall survival was also similar between the fulvestrant and anastrozole treatment arms (Pippen J et al 2003). Fulvestrant has received approval in 70 countries worldwide at this dose regimen.

However, evidence from a number of studies suggests that higher dose may be able to enhance efficacy further:

* Data from Study 0036 (Addo S et al, 2002) suggested that a dose-response relationship may exist. In female volunteers given a single intramuscular (i.m.) injection of fulvestrant (250mg, 125mg or placebo), there was a dose-dependent inhibition of ethinyloestradiol-induced endometrial thickening seen at Day 28.
* Results from short term exposure to fulvestrant in Studies 0002 (DeFriend D et al 1994) and 0018 (Robertson et al 2001) showed that expression of ER, progesterone receptor (PgR) and the cell proliferation-related antigen Ki67 are reduced in a dose-dependent manner.
* Data from Studies 0020 (Howell et al 2002) and 0021(Osborne CK et al 2002) suggested that a dose-response effect exists for fulvestrant. Fulvestrant 250mg was shown to be superior to fulvestrant 125mg, which was discontinued as it failed to meet minimum efficacy requirements.
* Evidence from pharmacokinetic modelling indicated that fulvestrant 500 mg dose regiment can achieve higher steady state plasma concentrations compared with fulvestrant 250mg and that steady state concentrations can be achieved earlier than with fulvestrant 250mg.
* Data from Study CONFIRM (A Di Leo et al 2009), a phase III randomised parallel-group trial, demonstrated that fulvestrant 500mg offers a statistically significant longer TTP compared with fulvestrant 250mg (median TTP: 6.5 months vs. 5.5 months; hazard ratio=0.80 [95% CI 0.68 to 0.94]; P=0.006), which seemed to be the consequence of an increase in the rate, and of a prolongation in duration, of disease stabilization. The 50% events overall survival analysis also seemed to favour fulvestrant 500mg, although statistical significance was not reached(hazard ratio=0.84 [95% CI 0.69 to 1.03]; P=0.091). The safety analysis did not raise any relevant concerns in relation to fulvestrant 500mg. Therefore, this study will compare Fulvestrant 500mg with fulvestrant 250mg in a Chinese population in order to understand the optimal dose for Chinese patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women defined as a woman who has stopped having menstrual periods
* Breast Cancer has continued to grow after having received treatment with an anti-estrogen hormonal treatment such as tamoxifen or an aromatase inhibitor
* Requiring hormonal treatment
* Oestrogen-receptor positive tumour
* Written informed consent to participate in the trial

Exclusion Criteria:

* Treatment with an investigational or non-approved drug within one month
* An existing serious disease, illness, or condition that will prevent participation or compliance with study procedures
* A history of allergies to any active or inactive ingredients of fulvestrant (i.e. castor oil)
* Treatment with more than one regimen of chemotherapy for advanced breast cancer
* Treatment with more than one regimen of hormonal treatment for advanced breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2011-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zefei Jiang, Principal Investigator — 307 Hospital of PLA; Yuri E Rukazenkov, Study Director — AstraZeneca
Locations (15):
- China (15):
  - Research Site, Beijing
  - Research Site, Chongqing
  - Research Site, Dalian
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Jiangsu
  - Research Site, Kunming
  - Research Site, Nanning
  - Research Site, Shandong
  - Research Site, Shanghai
  - Research Site, Shijiazhuang
  - Research Site, Taiyuan
  - Research Site, Tianjin

REFERENCES:
- See also: D6997L00021_CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=593&filename=D6997L00021_CSR_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The planned population size was 220 randomised patients. 249 patients were enrolled with 28 screen-failured patients and altogether 221 patients were randomised. The recuitment period of this study took 34 months, first subject in on 01 Mar 2011 and last subject in on 23 Dec 2013.
Pre-assignment Details: The Enrollment number in the protocol section means the number of patients enter the trial and receiving screening procedure, the number of participants Started in the Participant Flow module means the number of randomized patients and do not include screening failure patients.
Groups:
- Fulvestrant 500 mg: Fulvestrant 500 mg intramuscular (im) every 28 (± 3) days plus an additional 500 mg on Day 15 (± 3) of first month only
- Fulvestrant 250 mg: Fulvestrant 250 mg im every 28 (± 3) days
Period: Overall Study
Arm/Group | Fulvestrant 500 mg | Fulvestrant 250 mg
Started | 111 | 110
Received Study Treatment | 109 | 110
Completed | 75 | 72
Not Completed | 36 | 38
Not completed — Did not receive treatment | 2 | 0
Not completed — Ongoing treatment at data cut-off | 27 | 23
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 0 | 4
Not completed — Withdrawal by Subject | 7 | 10

BASELINE CHARACTERISTICS:
Population: The planned population size was 220 randomised patients and altogether 221 patients were randomised. Key demographic and baseline characteristics were balanced between the treatment groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fulvestrant 500 mg | Fulvestrant 250 mg | Total
Number analyzed (Participants) | 111 | 110 | 221
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (10.12) | 53.1 (10.22) | 53.3 (10.15)
Age, Customized [Number; unit: participants]
  <50 Years | 37 | 40 | 77
  ≥50 to <65 Years | 61 | 56 | 117
  ≥65 Years | 13 | 14 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 110 | 221
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants] — A PHASE III STUDY OF FULVESTRANT 500 MG VERSUS 250 MG IN POSTMENOPAUSAL CHINESE WOMEN WITH ADVANCED BREAST CANCER AND DISEASE PROGRESSION FOLLOWING FAILURE ON PRIOR ANTIESTROGEN OR AROMATASE INHIBITOR THERAPY
  Participants
    Asian | 111 | 110 | 221
Weight [Mean (Full Range); unit: kg] | 61.0 [35.0 to 85.0] | 60.5 [42.0 to 88.0] | 60.7 [35.0 to 88.0]
WHO Performance Status [Number; unit: participants]
  (0) Normal activity | 80 | 77 | 157
  (1) Restricted activity | 28 | 30 | 58
  (2) In bed ≤50% of the time | 3 | 3 | 6
Extent of disease at baseline [Number; unit: participants]
  Locally advanced breast cancer only | 1 | 1 | 2
  Metastatic disease | 110 | 109 | 219

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, or unequivocal progression of existing non-target lesions, or the appearance of new lesions, or death (by any cause in the absence of progression). The primary analysis for PFS was the log rank test stratified by last endocrine therapy received prior to fulvestrant (AO vs. AI). The treatment effect was estimated using the HR of 500 mg fulvestrant to 250 mg fulvestrant together with the corresponding 95% CI and p value.
Time Frame: 36 months
Population: FAS: all randomised patients and compared the treatment groups on the basis of randomised treatment, regardless of treatment actually received.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Fulvestrant 500 mg | Fulvestrant 250 mg
Number analyzed (Participants) | 111 | 110
months | 8.0 [2.8 to 16.6] | 4.0 [2.7 to 11.1]
Statistical Analysis 1: Comparison: Fulvestrant 500 mg vs Fulvestrant 250 mg; The results of this study would be considered to be consistent with that of the CONFIRM study if the hazard ratio (HR) point estimate for the treatment comparison was <1 (ie, it favoured fulvestrant 500 mg), without the requirement for the benefit of fulvestrant 500 mg to be statistically significant; Test type: Superiority or Other; p = 0.078, Log Rank — With a sample size of 220 randomised patients and 150 progression events, if treatment effect is consistent between ethnicities/the study populations, there is an 89% chance the HR <1; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.54 to 1.03]

2. Secondary Outcome: Objective Response Rate
Description: The ORR is defined as the proportion of all randomized patients with measurable disease at baseline who have a best objective tumour response of either CR or PR per RECIST v1.1.
Time Frame: 36 months
Population: Evaluable for Response Set, included all patients in the FAS with measurable disease at baseline.
Measure: Number; unit: patients
Arm/Group | Fulvestrant 500 mg | Fulvestrant 250 mg
Number analyzed (Participants) | 57 | 66
patients | 16 [5.36 to 11.04] | 11 [2.92 to 5.72]
Statistical Analysis 1: Comparison: Fulvestrant 500 mg vs Fulvestrant 250 mg; Test type: Superiority or Other; p = 0.107, Regression, Logistic; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.93 to 2.24]

3. Secondary Outcome: Clinical Benefit Rate
Description: A clinical benefit (CB) responder is defined as a patient having a best overall response of either CR, PR or SD for at least 24 weeks per RECIST v1.1. As tumour assessments can occur ± 2 weeks of the specified time point, the CBR is defined as the proportion of patients in the FAS who have CB ≥ 22 weeks (or 154 days).
Time Frame: 36 months
Population: FAS
Measure: Number; unit: patients
Arm/Group | Fulvestrant 500 mg | Fulvestrant 250 mg
Number analyzed (Participants) | 111 | 110
patients | 53 | 36
Statistical Analysis 1: Comparison: Fulvestrant 500 mg vs Fulvestrant 250 mg; Test type: Superiority or Other; p = 0.023, Regression, Logistic; Odds Ratio (OR) = 1.37, 95% CI 2-sided [1.04 to 1.80]

4. Secondary Outcome: Duration of Response
Description: Duration of response (DoR) will be evaluated only for patients who have an objective response, and is defined as the time from the date of first documentation of objective response (i.e., the initial visit at which CR or PR was recorded) until the date of disease progression or death due to any cause (whichever is earlier). The time of the initial response will be defined as the latest of the dates contributing towards the first visit response of PR or CR.
  Any patient who has not progressed or died by the date of DCO, or who has been lost to follow up, will be right-censored at the date of their last disease assessment.
Time Frame: 36 months
Population: Evaluable for Response Set
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Fulvestrant 500 mg | Fulvestrant 250 mg
Number analyzed (Participants) | 16 | 11
months | 16.6 [5.6 to NA] — The data is not available due to high percent (7/16, 43.75%) of patients censored. | 22.2 [10.8 to NA] — The data is not available due to high percent (8/11, 72.73%) of patients censored.

5. Secondary Outcome: Duration of Clinical Benefit
Description: Duration of clinical benefit (DoCB) will be evaluated only for patients who have CB, and is defined as the time from the date of randomisation until the date of disease progression or death from any cause, whichever is earlier.
  Any patient who has not progressed or died by the date of DCO or who has been lost to follow up will be right censored at the date of their last evaluable disease assessment.
Time Frame: 36 months
Population: FAS
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Fulvestrant 500 mg | Fulvestrant 250 mg
Number analyzed (Participants) | 53 | 36
months | 14.3 [11.0 to 25.0] | 13.8 [11.0 to NA] — The data is not available due to high percent (21/36, 58.33%) of patients censored.

ADVERSE EVENTS:
Time Frame: Adverse Events will be collected from time of signature of informed consent throughout the treatment period and up to 8 weeks after the last injection of study medication.
Arm/Group | Fulvestrant 500 mg | Fulvestrant 250 mg
Serious Adverse Events (participants affected / at risk) | 4/109 | 9/110
Other Adverse Events (participants affected / at risk) | 68/109 | 65/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant 500 mg (N=109) | Fulvestrant 250 mg (N=110)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 2
Lung infection (Infections and infestations) | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 0
Platelet count decreased (Investigations) | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant 500 mg (N=109) | Fulvestrant 250 mg (N=110)
INJECTION SITE REACTION (General disorders) | 12 | 13
INJECTION SITE PAIN (General disorders) | 8 | 10
FATIGUE (General disorders) | 9 | 7
NAUSEA (Gastrointestinal disorders) | 6 | 7
BACK PAIN (Musculoskeletal and connective tissue disorders) | 8 | 4
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 6
ANAEMIA (Blood and lymphatic system disorders) | 2 | 3
BONE MARROW FAILURE (Blood and lymphatic system disorders) | 2 | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 2
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1
HAEMOLYTIC URAEMIC SYNDROME (Blood and lymphatic system disorders) | 0 | 1
LYMPHADENITIS (Blood and lymphatic system disorders) | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1
PALPITATIONS (Cardiac disorders) | 1 | 2
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 0 | 1
SINUS TACHYCARDIA (Cardiac disorders) | 1 | 0
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 | 0
DEAFNESS UNILATERAL (Ear and labyrinth disorders) | 0 | 1
EAR PAIN (Ear and labyrinth disorders) | 1 | 0
TINNITUS (Ear and labyrinth disorders) | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 1 | 0
EYELID OEDEMA (Eye disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 4 | 2
DIARRHOEA (Gastrointestinal disorders) | 1 | 3
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 1
CONSTIPATION (Gastrointestinal disorders) | 2 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 | 1
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1
ASCITES (Gastrointestinal disorders) | 0 | 1
FAECES HARD (Gastrointestinal disorders) | 0 | 1
GASTRITIS (Gastrointestinal disorders) | 1 | 0
GINGIVAL PAIN (Gastrointestinal disorders) | 0 | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 1
MOUTH ULCERATION (Gastrointestinal disorders) | 1 | 0
TOOTHACHE (Gastrointestinal disorders) | 1 | 0
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 2 | 2
PYREXIA (General disorders) | 11 | 6
MALAISE (General disorders) | 3 | 2
OEDEMA PERIPHERAL (General disorders) | 2 | 2
INJECTION SITE PRURITUS (General disorders) | 1 | 2
ASTHENIA (General disorders) | 1 | 1
INJECTION SITE ANAESTHESIA (General disorders) | 1 | 1
INJECTION SITE MASS (General disorders) | 1 | 1
LOCAL SWELLING (General disorders) | 2 | 0
FACE OEDEMA (General disorders) | 0 | 1
INJECTION SITE INDURATION (General disorders) | 0 | 1
INJECTION SITE JOINT PAIN (General disorders) | 0 | 1
INJECTION SITE RASH (General disorders) | 1 | 0
INJECTION SITE SWELLING (General disorders) | 0 | 1
OEDEMA (General disorders) | 0 | 1
PAIN (General disorders) | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 3 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 2
LUNG INFECTION (Infections and infestations) | 1 | 2
URINARY TRACT INFECTION (Infections and infestations) | 1 | 1
ARTHRITIS BACTERIAL (Infections and infestations) | 0 | 1
BRONCHOPNEUMONIA (Infections and infestations) | 0 | 1
INFLUENZA (Infections and infestations) | 1 | 0
LARYNGITIS (Infections and infestations) | 1 | 0
LIP INFECTION (Infections and infestations) | 1 | 0
PHARYNGITIS (Infections and infestations) | 1 | 0
URETHRITIS (Infections and infestations) | 1 | 0
VIRAL RHINITIS (Infections and infestations) | 0 | 1
VULVITIS (Infections and infestations) | 1 | 0
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
INJECTION RELATED REACTION (Injury, poisoning and procedural complications) | 0 | 1
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 | 1
NEUTROPHIL COUNT DECREASED (Investigations) | 4 | 4
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 5 | 2
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 | 3
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 3 | 2
PLATELET COUNT DECREASED (Investigations) | 2 | 3
WEIGHT DECREASED (Investigations) | 1 | 1
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 | 0
BLOOD CREATININE INCREASED (Investigations) | 0 | 1
BLOOD FIBRINOGEN DECREASED (Investigations) | 0 | 1
ELECTROCARDIOGRAM ABNORMAL (Investigations) | 1 | 0
HAEMOGLOBIN DECREASED (Investigations) | 1 | 0
HEPATIC ENZYME INCREASED (Investigations) | 1 | 0
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 4 | 3
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 1
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 4 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 | 1
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 1
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 | 1
HEADACHE (Nervous system disorders) | 7 | 4
DIZZINESS (Nervous system disorders) | 1 | 2
CEREBRAL INFARCTION (Nervous system disorders) | 1 | 0
EPILEPSY (Nervous system disorders) | 1 | 0
FACIAL NERVE DISORDER (Nervous system disorders) | 1 | 0
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 | 1
HYPERSOMNIA (Nervous system disorders) | 0 | 1
HYPOAESTHESIA (Nervous system disorders) | 1 | 0
INSOMNIA (Psychiatric disorders) | 2 | 1
MENOPAUSAL DEPRESSION (Psychiatric disorders) | 1 | 0
RESTLESSNESS (Psychiatric disorders) | 1 | 0
BREAST SWELLING (Reproductive system and breast disorders) | 1 | 0
MENOPAUSAL SYMPTOMS (Reproductive system and breast disorders) | 0 | 1
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 4 | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 2
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
LARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 3 | 1
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 1 | 0
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 | 0
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 1
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 | 1
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 1
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 1 | 0
SKIN MASS (Skin and subcutaneous tissue disorders) | 0 | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 1 | 0
HYPERTENSION (Vascular disorders) | 3 | 1
HOT FLUSH (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
China CONFIRM Study was planned as a bridge study to the CONFIRM Study and therefore was not formally powered to detect a statistically significant difference between two treatment groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No